CLINICAL TRIAL: NCT07203833
Title: Diagnostic and Prognostic Evaluation of Vasorin During Septic Shock
Acronym: VASO-DIAG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2025_843_0152
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Vasorin; Septic Shock; Shock; Biomarker; Infection
Keywords: Septic shock; vasorin; Shock; Biomarker; Infection
MeSH Terms: conditions — Shock, Septic; Shock; Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- in septic shock (infection) (Experimental)
  Interventions: Biological: blood sample
- in shock without sepsis (without infection) (Active Comparator)
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — blood sample in order to measure the concentrations of circulating Vasn

SUMMARY:
Septic shock is the most severe form of infection. Currently, an early specific biomarker for septic shock is needed. Remember that shock situations are numerous, not only septic (eg hemorrhagic, cardiogenic...), and also accompanied by a severe pro-inflammatory state that it is sometimes difficult to distinguish from a septic state. Procalcitonin (PCT) is the most studied biomarker but still lacks sensitivity (77%) and specificity (79%). The investigators hypothesize that the Vasn could become this potential new biomarker and would allow a better diagnosis and thus the need or not to treat patients with antibiotics. The laboratory studies suggest a link between Vasn and septic shock. The goal of this project is to measure and compare plasma Vasn concentrations in 2 groups of patients = group 1: septic shock versus group 2: non-septic shock. Briefly, shock is defined as low blood pressure requiring vasopressor agents with confirmed infection (group 1) or without suspected infection such as patients admitted in intensive care unit post cardiac surgery with CBP (group 2). The investigators will also assess patient 28-day mortality to identify Vasn as a potential prognostic biomarker.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years.
* Patients admitted for less than 24 hours in intensive care unit of the CHU Amiens Picardie.
* Group 1: patients with septic shock defined by sepsis with 2 mmol/l Lactates, requiring vasopressors to maintain mean blood pressure at 65 mmHg (despite adequate vascular filling) in the presence of fever (T°>38.3) with a documented or suspected infection
* Group 2: patients with a shock defined by arterial hypotension requiring the use of vasopressors with 2 mmol/l Lactates but without suspected infection and apyrexie (T°<38°). For example: vasoplegia post cardiac surgery with CBP or cardiogenic shock or hemorrhagic shock

Exclusion Criteria:

* Pregnant women
* Group 1 : No evidence of suspected or documented infection
* Group 2 : Presence of fever and/or suspected infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-10-19 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Vasn plasma concentration at D0 for each group | day 0
Vasn plasma concentration in each group | day 1
Vasn plasma concentration in each group | day 3
Correlation between Vasn plasma concentration and noradrenaline dose peak in each group | day 0
Correlation between Vasn plasma concentration and noradrenaline dose peak in each group | day 1
Correlation between Vasn plasma concentration and noradrenaline dose peak in each group | day 3
Correlation between Vasn plasma concentration and occurrence of an IRA (KDIGO score) in each group | day 0
Correlation between Vasn plasma concentration and occurrence of an IRA (KDIGO score) in each group | day 1
Correlation between Vasn plasma concentration and occurrence of an IRA (KDIGO score) in each group | day 3
Correlation between Vasn plasma concentration and coagulation marker concentration in each group | day 0
  coagulation marker are TF, platelet count, TP, TCA, Factor V, fibrinogen, D-dimers
Correlation between Vasn plasma concentration and coagulation marker concentration in each group | day 1
  coagulation marker are TF, platelet count, TP, TCA, Factor V, fibrinogen, D-dimers
Correlation between Vasn plasma concentration and coagulation marker concentration in each group | day 3
  coagulation marker are TF, platelet count, TP, TCA, Factor V, fibrinogen, D-dimers
Correlation between Vasn plasma concentration and SOFA score at admission in each group | day 0
Correlation between Vasn plasma concentration and SOFA score at admission in each group | day 1
Correlation between Vasn plasma concentration and mortality in each group | day 3
Correlation between Vasn plasma concentration and SOFA score at admission in each group | day 3
Correlation between Vasn plasma concentration and mortality in each group | day 0
Correlation between Vasn plasma concentration and mortality in each group | day 1
Correlation between Vasn plasma concentration and length of hospitalization in each group | day 1
Correlation between Vasn plasma concentration and length of hospitalization in each group | day 0
Correlation between Vasn plasma concentration and length of hospitalization in each group | day 3
Correlation between Vasn plasma concentration and plasma level of procalcitonin in each group | day 0
Correlation between Vasn plasma concentration and plasma level of procalcitonin in each group | day 1
Correlation between Vasn plasma concentration and plasma level of procalcitonin in each group | day 3

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No